CLINICAL TRIAL: NCT01045044
Title: Magnetic Resonance Imaging of Tumor Response and Cognitive Impairment in Breast Cancer Patients Undergoing Anthracycline-based Systemic Chemotherapy
Brief Title: Magnetic Resonance Imaging (MRI) of Tumor Response and Cognitive Impairment in Breast Cancer Patients Undergoing Chemotherapy
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: Kettering Health Network (Other)
Responsible Party: Jason Parker, PhD, Kettering Health Network Innovation Center
Other Study IDs: KHNIC-P09-004
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Magnetic Resonance Imaging; Anthracycline based systemic chemotherapy; Tumor response; Cognitive Impairment; Chemo Brain
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breast cancer, chemotherapy: Up to 15 women with breast cancer who are to undergo systemic anthracycline based chemotherapy.
- Normal control: Up to 15 normal, healthy women.

SUMMARY:
We will use magnetic resonance imaging (MRI) to investigate tumor changes in women with breast cancer who are receiving anthracycline-based systemic chemotherapy. We will also use MRI and cognitive tests to study the possible effects of chemotherapy on the brains of these women. The results will be compared to a control group of normal healthy women. We will try to determine if MRI can be used to predict tumor response and cognitive changes related to the chemotherapy.

DETAILED DESCRIPTION:
In this work we will utilize conventional magnetic resonance imaging as well as a set of advanced magnetic resonance imaging tools to investigate changes in tumor physiology and the human brain resulting from anthracycline-based systemic chemotherapy. We will recruit up to 15 subjects diagnosed with breast cancer and preparing for an anthracycline-based systemic chemotherapy regimen. Each subject will undergo the set of MR imaging tools before therapy, after one therapy session, after four therapy sessions, and at the conclusion of therapy. Conventional MRI methods will be used to quantify tumor-response to chemotherapy for each subject. A control group of up to 15 normal subjects will also be recruited and will undergo MR brain imaging twice with a gap of 6 months between scans. All subjects will also undergo a battery of neuropsychological tests at each imaging session. The results of the neuropsychological tests will be used to quantify cognitive changes for each subject. A final analysis will determine if the advanced MR modalities can be used to predict the response of tumors or human cognition to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Adenocarcinoma(ER+ve, PR+ve)
* Prescribed, but not yet begun, anthracycline based systemic chemotherapy
* Not prescribed Avastin
* Able to read and write in English
* Have signed informed consent

Exclusion Criteria:

* Diagnosed psychiatric disorder
* Conditions that would preclude MRI (Pacemaker, metal objects in body, claustrophobia, pregnancy, etc.)
* Serious, unstable medical or mental illness
* Medical contraindication to any study procedure
* Current alcohol or other substance use disorder (excluding nicotine)
* Have not read and signed informed consent, or do not understand its contents

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer cohort will be patients of Medical Oncology Hematology Associates Inc., Dayton, OH
  Normal controls will be recruited from Kettering College of Medical Arts and the Kettering Health Network.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Parker, PhD, Principal Investigator — Kettering Health Network
Locations (2):
- United States (2):
  - Medical Oncology Hematology Associates, Inc, Dayton, Ohio
  - Innovation Center, Kettering Health Network, Kettering, Ohio